CLINICAL TRIAL: NCT04102683
Title: The Effects of Therapeutic Recreation Activities on Emotional Adjustment of Individuals With Intellectual Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ezgi Ertüzün, Associate professor, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 123456
Record Dates: First submitted 2019-09-16; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Emotional Adjustment; Intellectual Disability
Keywords: Game; Therapeutic Recreation; Intellectual Disability
MeSH Terms: conditions — Intellectual Disability

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The experimental recreation program, which consisted of two sessions per week and lasted approximately 1 hour each session, lasted for 8 weeks between March 2019 and May 2019 for the adolescents in the experimental group. The Therapeutic Recreation Activity Program, which consists of 16 sessions, is organized according to the self-determination and entertainment development model. This model aims to provide individual development and prosperity by creating an entertaining environment with therapeutic recreation. According to the degree of enjoyment, activity improves freedom of choice, preferences and ability to express oneself. Pleasure is a feeling that the participant feels deeply during therapeutic recreation. Provides entertainment experience. Pleasure increases individual motivation to participate, as well as making the best use of physical, social and emotional conditions.
  Interventions: Behavioral: Therapeutic recreation activity program
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Therapeutic recreation activity program — The experimental recreation program, which consisted of two sessions per week and lasted approximately 1 hour each session, lasted for 8 weeks between March 2019 and May 2019 for the adolescents in the experimental group. The Therapeutic Recreation Activity Program, which consists of 16 sessions, is organized according to the self-determination and entertainment development model. This model aims to provide individual development and prosperity by creating an entertaining environment with therapeutic recreation. According to the degree of enjoyment, activity improves freedom of choice, preferences and ability to express oneself. Pleasure is a feeling that the participant feels deeply during therapeutic recreation. Provides entertainment experience. Pleasure increases individual motivation to participate, as well as making the best use of physical, social and emotional conditions.
  Arms: Intervention Group

SUMMARY:
The aim of this study was to determine the effect of Therapeutic Recreation Activities on Emotional Adjustment of Adolescents With Intellactual Disabilities. The research was carried out at Meram Melike Hatun Special Education Vocational School in Konya. The study took place between March 2019 and May 2019. The parents of the participants who participated in the study consisted of the experimental group (n = 17) and the remaining parents (n = 17) formed the control group and the sample group (n = 34). The personal information form which measures demographic characteristics developed by the researchers according to the literature, and Hacettepe Emotional Adjustment Scale were used. Data were analyzed in SPSS 22 program. According to Kolmogorov-Smirnov Z test, sample group was not normal. For this reason, non-parametric tests were performed. In descriptive data, the mean, number, percentage will be used; Comparative statistics were made according to the assumptions of non-parametric test (Wilcoxon test, Mann Whitney U test). Therapeutic Recreation Activities was applied as total of 16 sessions, consisting of two sessions per week and each session lasting about 1 hour. The program was implemented by researcher.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Having a physical disability,
* Having Down syndrome

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Mental adjustment scale score level | through study completion, an average of 1 year
  The scale, developed by Gökler and Öktem in 1985 (Kaner et al. 2012), consists of 32 items including psychological symptoms that may occur in every child. For each item, there are "None", "Some", "Many" options; scoring, 0, 1, 2 points, which are the equivalents of these options, are added to the scale. Single-digit items indicate neurotic problems and double-digit items indicate behavioral problems. The points up to Article 25 are added to the total scale. If a score of 13 or higher is obtained, it is said that there is a mental problem. Psychological Adjustment Scale; In order to determine the level of psychological adjustment of the participants, Neurotic Problems (12 items), Behavioral Problems (12 items) and Other behavior problems (7 items) included three factors. The internal consistency coefficient of this study was α = .80 for preliminary measurements; and .81 for the last measurements

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided